CLINICAL TRIAL: NCT04515628
Title: An Open-Label, Single-Sequence Crossover, Drug-Drug Interaction Study to Assess the Effect of Steady-State Branebrutinib on the Pharmacokinetics of Rosuvastatin in Healthy Participants
Brief Title: Study to Assess the Effect of Branebrutinib on the Drug Levels of Rosuvastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM014-032
Record Dates: First submitted 2020-08-14; First posted 2020-08-17 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Rosuvastatin Calcium; branebrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Period A: Rosuvastatin (Experimental)
  Interventions: Drug: Rosuvastatin
- Period B: Branebrutinib (Experimental)
  Interventions: Drug: Branebrutinib
- Period C: Branebrutinib + Rosuvastatin and Branebrutinib (Experimental)
  Interventions: Drug: Rosuvastatin; Drug: Branebrutinib
- Period D: Branebrutinib (Experimental)
  Interventions: Drug: Branebrutinib

INTERVENTIONS:
Drug: Rosuvastatin — Specified dose on specified days
  Arms: Period A: Rosuvastatin; Period C: Branebrutinib + Rosuvastatin and Branebrutinib
Drug: Branebrutinib — Specified dose on specified days
  Arms: Period B: Branebrutinib; Period C: Branebrutinib + Rosuvastatin and Branebrutinib; Period D: Branebrutinib

SUMMARY:
The purpose of this study is to examine the interaction of branebrutinib with rosuvastatin. Rosuvastatin is a substrate of the breast cancer resistance protein (BCRP) transporter, which has a drug level profile that can be markedly altered by coadministration of known inhibitors of the BCRP transporter. With widespread use of statins as cholesterol-lowering agents, rosuvastatin is also a likely concomitant drug for participants who would potentially be treated with branebrutinib.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participant, as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations by investigator
* Body mass index (BMI) of 18.0 kg/m2 to 32.0 kg/m2, inclusive, as measured at screening visit
* Women and men must agree to follow specific methods of contraception, if applicable, while participating in the trial

Exclusion Criteria:

* Women who are of childbearing potential
* Women who are pregnant or breastfeeding
* Any significant acute or chronic medical illness that presents a potential risk to the participant in the opinion of the investigator and/or may compromise the objectives of the study, including a history of or active liver disease
* Any other sound medical, psychiatric, and/or social reason as determined by the investigator

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-02 (Actual); Primary Completion 2020-10-18 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of rosuvastatin | Up to 6 days
Maximum observed plasma concentration (Cmax) of rosuvastatin when coadministered with branebrutinib | Day 13
Area under the concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of rosuvastatin | Up to 6 days
Area under the concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of rosuvastatin when coadministered with branebrutinib | Day 13
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] of rosuvastatin | Up to 6 days
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] of rosuvastatin when coadministered with branebrutinib | Day 13

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 33 days
Incidence of Serious Adverse Events (SAEs) | Up to 77 days
Incidence of AEs leading to discontinuation | Up to 33 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 54 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 54 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 54 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 54 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to 54 days
  PR interval: The time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QRS interval | Up to 54 days
  QRS interval: A combination of the Q wave, R wave and S wave, the "QRS complex" represents ventricular depolarization
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QT interval | Up to 54 days
  QT interval: Measured from the beginning of the QRS complex to the end of the T wave
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QTcF interval | Up to 54 days
  QTcF interval: Corrected QT interval using Fridericia's formula (QTcF)
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 53 days
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 53 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 53 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON (LPRA) - Salt Lake, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm